CLINICAL TRIAL: NCT04329143
Title: Post-Cholecystectomy Gall Bladder Remnant and Cystic Duct Stump Stone: Surgical Pitfalls, Causes of Occurrence and Completion Cholecystectomy (Open Vs Laparoscopic) as a Safe Surgical Option of Treatment
Brief Title: Post-Cholecystectomy Gall Bladder Remnant and Cystic Duct Stump Stone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer Alsaied Alnaimy, assistant professour, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: cystic duct stump stone
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-03

CONDITIONS: Laparocele
Keywords: Post cholecystectomy; Stump; stone
MeSH Terms: conditions — Postcholecystectomy Syndrome; Calculi

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- open completion cholecystectomy (Active Comparator): open completion cholecystectomy for cystic duct stump stone
  Interventions: Procedure: open completion cholecystectomy
- laparoscopic completion cholecystectomy (Active Comparator): lap completion cholecystectomy for cystic duct stump stone
  Interventions: Procedure: lap completion cholecystectomy

INTERVENTIONS:
Procedure: open completion cholecystectomy — open excision of cystic duct remnant
  Arms: open completion cholecystectomy
Procedure: lap completion cholecystectomy — lap excision of cystic duct stone
  Arms: laparoscopic completion cholecystectomy

SUMMARY:
Introduction: cholecystectomy relieves pre-surgical symptoms of gallbladder disease. The persistence of symptoms was recorded in 10 - 20% of cases. Residual gall bladder/cystic duct stump stone is one of the most important cause.

Aim: to compare between open and laparoscopic completion cholecystectomy of gall bladder remnant and cystic duct stump syndrome as regard short and long term outcome.

Methods: This prospective study was conducted on 20 cases with residual GB/cystic duct stump stone. The diagnosis was guided by ultrasound and magnetic resonance cholangio-pancreatography. All cases were managed by using completion cholecystectomy - either open or laparoscopic. All preoperative, operative, and postoperative data were collected...

DETAILED DESCRIPTION:
The incidence of gall bladder and cystic duct stump stones has been reported to be 5% of patients after urgent cholecystectomy, and it is rare after elective operations . The incidence of incomplete gallbladder removal following laparoscopic cholecystectomy is 13.3% . Partial cholecystectomy may be resorted to in many conditions such as difficult dissection in Calot's triangle that can be hazardous to common bile duct and/or blood vessels. In such cases, many surgeons leave a part of the gall bladder in the manner described by author after removing all stones from the remaining cuff of the gallbladder To prevent the incidence of gallbladder remnant/cystic duct stump calculi, the cystic duct should be fully skeletonized till 1 cm from the common bile duct. Stones in the cystic duct should be milked back to the gallbladder before clipping Routine use of intraoperative cholangiography is not a must but when used it can be useful in detecting calculi in the cystic duct The diagnosis of cystic duct stump syndrome is always into the dilemma of post cholecystectomy syndromes and leads to delayed diagnosis. Cystic duct stump syndrome may be misdiagnosed with reflux esophagitis, peptic ulceration, irritable bowel syndrome or chronic pancreatitis hepatitis, mesenteric ischemia, diverticulitis, and organic or motor intestinal disorders.

The imaging approach to post cholecystectomy syndrome includes ultrasonography, computed tomography (CT) scan, endoscopic retrograde cholangiopancreatography (ERCP), and magnetic resonance cholangiopancreatography (MRCP).

The purpose of this study is to emphasis that laparoscopic completion cholecystectomy is the best surgical option for cystic duct stump and gall bladder remnant syndrome as regard safety to the patients...

There may be gender specific risk factor for developing post-cholecystectomy syndrome, in present study; the incidence was 70% in females (14 cases) compared to 30% in males (6 cases). This higher incidence in females was also reported , whom stated that the male to female ratio was 1:1.45.

The symptoms of gall bladder syndrome may be nil or they can present with acute symptoms (biliary colic, acute cholecystitis or acute pancreatitis) or chronic symptoms (persistent right upper quadrant discomfort or pain, food intolerance, nausea or jaundice). The persistence of symptoms after cholecystectomy points to the possibility of a gallbladder remnant, especially when coupled with radiation of pain to the shoulder, food intolerance, nausea or jaundice . abdominal pain and persistent dyspepsia as the commonest presentation were stated by other study , while , reported that patients was referred to their institution without persistent symptoms after cholecystectomy .In the present study, most cases presented with right hypochondrial pain (18 cases) and asymptomatic cases are 2 cases and discovered accidently by ultrasonography for other unrelated symptoms.

ELIGIBILITY:
Inclusion Criteria:

* • Age: 30-50

  * Both sex
  * Previous cholecystectomy(open or laparoscopic)
  * With or without common bile duct stone.
  * Symptomatic or

Exclusion Criteria:

* • 1-patients unfit for surgery

  * 2-patient refused surgery.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
postoperative pain severity on visual analogue score | 2 weeks
  assessement of pain severity after operation in record of 10

SECONDARY OUTCOMES:
intraoperative time in minutes | 2 hours
  assessement of time in the operation in minutes

CONTACTS AND LOCATIONS:
Overall Officials: tamer A. alnaimy, MD, Principal Investigator — Zagazig University

IPD SHARING:
Plan to Share IPD: No